CLINICAL TRIAL: NCT07020286
Title: Prince of Wales Hospital Structural Heart Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Principle investigator, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: 2024.199
Record Dates: First submitted 2024-11-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Structural Heart Abnormality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject: Structural heart intervensions
  Interventions: Procedure: Structural heart interventions

INTERVENTIONS:
Procedure: Structural heart interventions — The study allows us to understand the trend of transcatheter interventions in structural heart disease, clinical outcomes and allows the comparison of the outcomes of structural heart interventions to medical therapy and surgery at PWH, and to HA hospitals.

SUMMARY:
Structural heart disease refers to a group of cardiac defects other than coronary artery disease. Structural heart intervention is a rapidly growing field in cardiology. In the past decade, there has been paradigm shift in the management of structural heart disease from conventional open-heart surgery to transcatheter interventions. With increasing evidence supporting structural heart interventions including transcatheter aortic valve implantation or transcatheter edge to edge repair, there has important updates in recent guidelines in treating structural heart disease. Besides, new device innovations bloomed over the past few years and had expanded the possible treatment options for high surgical risk patients. Some breakthrough devices had been approved recently by the US Food and Drug Administration and some other devices are occasionally used on compassionate ground. However, there has been lack of data in structural heart interventions in Asia Pacific regions outside Japan [8]. In this study, we would like to analyze the epidemiological trends, patient characteristics, procedural outcomes and clinical outcomes of structural heart interventions, and compare them with historical cohorts, matched cohort receiving medical therapy and matched cohort receiving open heart surgeries.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing structural heart interventions at the Prince of Wales Hospital

Exclusion Criteria:

* Patients that are not able to consent.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: There is approximately 250 cases of structural heart intervention cases performed in 2023. The numbers are stable in the past 3 years. The dropout rate around 1-2% as reflected from other registry studies. Therefore, there would be around 1000 cases to be recruited during our 4 year recruitment period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Procedural success rate | Post-procedure until 1 year post OP
  Procedural success rate
Procedural safety endpoints | Post-procedure until 1 year post OP
  Rate of vascular complication in enrolled subjects , ,
Procedural safety endpoints | Post-procedure until 1 year post OP
  Rate of myocardial infarction in enrolled subjects
Procedural safety endpoints | Post-procedure until 1 year post OP
  Rate of stroke in enrolled subjects
Procedural safety endpoints | Post-procedure until 1 year post OP
  Rate of cardiac perforation in enrolled subjects
Procedural safety endpoints | Post-procedure until 1 year post OP
  Rate of device embolization in enrolled subjects
Procedural safety endpoints | Post-procedure until 1 year post OP
  Rate of death in enrolled subjects
Procedural safety endpoints | Post-procedure until 1 year post OP
  Rate of conversion to open heart surgery in enrolled subjects

SECONDARY OUTCOMES:
Clinical outcome | 3 months
  NTproBNP at 3 months
Clinical outcome | 3 months
  NYHA class at 3 months
Clinical outcome | 12 months
  NTproBNP at 12 months
Clinical outcome | 12 months
  NYHA class at 12 months
Echocardiogram outcome | 3 months
  peri-device leak at post-OP 3 months compared with baseline
Echocardiogram outcome | 3 months
  LVEF at post-OP 3 months compared with baseline
Echocardiogram outcome | 3 months
  Valve residual regurgitation at post-OP 3 months compared with post-OP
Echocardiogram outcome | 3 months
  Degree of Valve stenosis at post-OP 3 months compared with baseline
Echocardiogram outcome | 12 months
  Degree of Valve stenosis at post-OP 12 months compared with baseline
Echocardiogram outcome | 12 months
  Peri-device leak at post-OP 12 months
Echocardiogram outcome | 12 months
  LVEF at post-OP 12 months compared with baseline
Echocardiogram outcome | 12 months
  valve residual regurgitation at post-OP 12 months compared with baseline
Clinical outcome | 12 months
  NYHA class comparison with matched historical cohort at PWH
  * Clinical outcome comparison with medical therapy cohort at PWH
  * Clinical outcome comparison with surgical cohort at PWH
  * Clinical outcome comparison with matched cohort at HA
Clinical outcome | 12 months
  NTproBNP comparison with matched historical cohort at PWH
  * Clinical outcome comparison with medical therapy cohort at PWH
  * Clinical outcome comparison with surgical cohort at PWH
  * Clinical outcome comparison with matched cohort at HA

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Xu, Research Nurse, Study Director — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD